CLINICAL TRIAL: NCT06907576
Title: Comparison of Labor Characteristics and Maternal-Neonatal Outcomes in Induced Labor Between Women With Gestational Hypertension/Mild Preeclampsia and Normotensive Controls
Brief Title: Labor Characteristics and Outcomes in Women With Gestational Hypertension or Preeclampsia Who Underwent Labor Induction
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2025-07-209
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Gestational Hypertension; Mild Pre-eclampsia
Keywords: induction of labor; gestational hypertension; mild pre-eclampsia
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- the HDP group: The pregnant women had combined with gestational hypertension or mild pre-eclampsia.
- the normotensive pregnancies group

SUMMARY:
Comparison of Labor Characteristics and Maternal-Neonatal Outcomes in Induced Labor Between Women with Gestational Hypertension/Mild Preeclampsia and Normotensive Controls

DETAILED DESCRIPTION:
The American College of Obstetricians and Gynecologists (ACOG) recommends that women with gestational hypertension or preeclampsia without severe features at or beyond 37 weeks of gestation are usually managed by scheduled induction of labor (IOL). Occasionally, normal pregnant women request elective induction of labor because of a perceived decrease in fetal movements in the presence of normal findings in fetal heart rate monitoring. However, there is limited information available to compare labor induction outcomes between patients with gestational hypertension or mild-preeclampsia and those with normal pregnancies. In addition, no studies have analyzed the characteristics and interventions of labor in hypertensive patients with induction of labor who undergone vaginal birth. Therefore, the purpose of this project was to investigate the differences of labor characteristics and maternal-neonatal outcomes with induction of labour (IOL) between pregnant women with gestational hypertension or mild pre-eclampsia and those with normotensive pregnancies, providing clinical references of intrapartum management for women with gestational hypertension or mild pre-eclampsia.

Our results showed that women with hypertensive pregnancies had higher rates of cesarean delivery due to failed induction compared to normotensive pregnancies. However, no significant differences were observed in induced labor characteristics, intrapartum interventions, and maternal-neonatal complications between women with gestational hypertension or mild pre-eclampsia and those with normotensive pregnancies. Parity, bishop score, birth weight, and the hypertensive disorders of pregnancy were independently and significantly associated with an increased risk of cesarean section following induction. Consequently, these findings could provide evidence for the intrapartum management of labor induction in women with gestational hypertension or mild pre-eclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing an induction of labor at term (37-42 weeks) who gave birth to a live born, non-anomalous singleton in cephalic presentation, as well as women aged 18-35 years old

Exclusion Criteria:

* Women with pregnancy complications including diabetes mellitus, intrahe-patic cholestasis of pregnancy, placenta previa, placental abruption, oligohydramnios, and polyhydramnios, previous caesarean births, fetal birth weight of ≥4.0 kg, severe preeclampsia, chronic hypertension, prepregnancy hypothyroidism and hyperthyroidism, renal system disease, nutritional deficiency, immune system disease, hematological system diseases, and prepregnancy thrombocytopenia. Women were also excluded if clinical data were incomplete.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This cohort study enrolled 425 pregnant women who underwent IOL, and they were divided into two groups: the HDP group and the normotensive pregnancies group.
Sampling Method: Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
the rate of cesarean delivery | 35 weeks to 40 weeks gestation
  pregnant outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ying Hua, Study Director — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- department of obstetrics of Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China